CLINICAL TRIAL: NCT00744991
Title: A Phase 2, Open-Label, Multicenter Study of Single-Agent Enzastaurin in Patients With Relapsed Cutaneous T-Cell Lymphoma
Brief Title: A Study for Participants With Relapsed Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11496; H6Q-MC-JCCB (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Cutaneous T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzastaurin (Experimental): Open Label
  Interventions: Drug: Enzastaurin

INTERVENTIONS:
Drug: Enzastaurin — 1125 milligrams (mg) loading dose then 500 mg, oral, daily, until disease progression
  Other Names: LY317615

SUMMARY:
The purpose of the study is to determine the efficacy and safety of enzastaurin in participants with Cutaneous T-Cell Lymphoma (CTCL) who failed prior therapies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed mycosis fungoides or Sezary Syndrome.
* Stage IB to IVB disease at screening.
* Recurrent or refractory disease after at least 1 prior systemic therapy.
* Have adequate organ function defined as:

  * Hepatic: total bilirubin ≤1.5 times the upper limit of normal (ULN); alanine transaminase/aspartate transaminase (ALT/AST) ≤2.5 times the ULN.
  * Renal: serum creatinine ≤1.5 times the ULN.
  * Adequate bone marrow reserve: platelets ≥75 * 10^9/Liters (L); absolute neutrophil count (ANC) ≥1.0 * 10^9/L.
* At least 30 days must have passed since other treatment for CTCL.

Exclusion Criteria:

* Receiving concurrent treatment for CTCL.
* Unable to swallow tablets.
* Receiving high potency oral or topical steroids. Low potency oral steroid may be permitted in participants who have been on a stable dose for at least 4 weeks prior to screening. Oral or topical antihistamine is allowed.
* Unable to discontinue use of carbamazepine, phenobarbital, or phenytoin.
* Have a serious concomitant systemic disorder or Human Immunodeficiency Virus (HIV).
* Have a serious cardiac condition such as myocardial infarction within past 6 months, angina, or heart disease as defined by the New York Heart Association (NYHA) Class III or IV.
* Have electrocardiogram (ECG) abnormalities.
* Are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- United States (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stanford, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas

REFERENCES:
- [Derived] Querfeld C, Kuzel TM, Kim YH, Porcu P, Duvic M, Musiek A, Rook AH, Mark LA, Pinter-Brown L, Hamid O, Lin B, Bian Y, Boye M, Day JM, Rosen ST. Multicenter phase II trial of enzastaurin in patients with relapsed or refractory advanced cutaneous T-cell lymphoma. Leuk Lymphoma. 2011 Aug;52(8):1474-80. doi: 10.3109/10428194.2011.572265. Epub 2011 Jun 8. PMID 21649541
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study had 2 stages. Stage 2 would occur if the minimum level of efficacy (confirmed complete or partial anti-tumor response) was observed in Stage 1. The study was considered complete at the end of Stage 1.
Groups:
- Enzastaurin: Enzastaurin 1125 milligrams (mg) loading dose (total 9 tablets; three 125-mg tablets administered orally 3 times) on Day 1 followed by 500 mg enzastaurin (total 4 tablets; two 125-mg tablets administered orally twice daily) with a minimum of 8 hours between the 2 doses starting on Day 2 until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
Period: Overall Study
Arm/Group | Enzastaurin
Started | 25
Received at Least 1 Dose | 25
Completed | 0
Not Completed | 25
Not completed — Progressive Disease | 11
Not completed — Withdrawal by Subject | 8
Not completed — Physician Decision | 3
Not completed — Adverse Event | 2
Not completed — Protocol Entry Criteria Unmet | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug.
Arm/Group | Enzastaurin
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 64 [26 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 18
  African | 4
  Hispanic | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Number of Participants with Cutaneous T-Cell Lymphoma (CTCL) Variant [Count of Participants; unit: Participants] — Mycosis Fungoides (MF) and Sezary Syndrome (SS) are the common types of Cutaneous T-Cell Lymphomas.
  Participants
    Mycosis Fungoides (MF) | 19
    Sezary Syndrome (SS) | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Complete Response (CR) or Partial Response (PR) Among Mycosis Fungoides (MF) and Sezary Syndrome (SS) Participants (Response Rate)
Description: Response rate is percentage of participants with confirmed CR or PR as per modified Severity-Weighted Assessment Tool (mSWAT) for MF group; mSWAT and Sezary count for SS group. mSWAT is a weighted sum of percent (%) of total body surface area attributed to skin lesions which yield a mSWAT score [0 (unaffected) to 400 (severely affected)] transformed into responses. As per mSWAT (CR: No detectable malignant disease for ≥4 weeks; PR: ≥50% mSWAT score reduction from baseline). Sezary cells percentage in lymphocytes measured using flow cytometry. As per Sezary count (CR: Sezary cells <5%; PR: ≥50% reduction in Sezary cells from baseline). Response rate is calculated as total number of participants with CR or PR from the start of study treatment until PD or recurrence divided by the number of participants treated, then multiplied by 100.
Time Frame: Baseline to measured Progressive Disease (PD) [up to 9 cycles (28-day cycles)]
Population: All participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Mycosis Fungoides (MF): Participants with histologically confirmed MF received enzastaurin 1125 milligrams (mg) loading dose (total 9 tablets; three 125-mg tablets administered orally 3 times) on Day 1 followed by 500 mg enzastaurin (total 4 tablets; two 125-mg tablets administered orally twice daily) with a minimum of 8 hours between the 2 doses starting on Day 2 until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- Sezary Syndrome (SS): Participants with histologically confirmed SS received enzastaurin 1125 mg loading dose (total 9 tablets; three 125-mg tablets administered orally 3 times) on Day 1 followed by 500 mg enzastaurin (total 4 tablets; two 125-mg tablets administered orally twice daily) with a minimum of 8 hours between the 2 doses starting on Day 2 until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
Arm/Group | Mycosis Fungoides (MF) | Sezary Syndrome (SS)
Number analyzed (Participants) | 19 | 6
percentage of participants
  Partial Response (PR) | 5.3 [0.1 to 26.0] | 0 [0 to 0]
  Complete Response (CR) | 0 [0 to 0] | 0 [0 to 0]

2. Secondary Outcome: Duration of Response for Responding Participants
Description: Time from first confirmed response [Complete Response (CR) or Partial Response (PR)] until Progressive Disease (PD) as per mSWAT for MF group; mSWAT and Sezary count for SS group. mSWAT: weighted sum of percent (%) of total body surface area attributed to skin lesions; scores [0 (unaffected) to 400 (severely affected)] transformed into responses. As per mSWAT (CR: No detectable malignant disease for ≥4 weeks; PR: ≥50% reduction in mSWAT score from baseline; PD: ≥25% of mSWAT score from nadir). Sezary cells percentage in lymphocytes measured using flow cytometry. As per Sezary count (CR: Sezary cells <5%; PR: ≥50% reduction in Sezary cells from baseline; PD: ≥40% of Sezary cells from nadir). Responders or those who died without PD were censored at date of last progression-free disease assessment. Responders who received subsequent systemic anticancer therapy were censored at date of last progression-free disease assessment prior to post-discontinuation therapy.
Time Frame: Time of response to PD [up to 9 cycles (28-day cycles)]
Population: Participants with confirmed response (CR or PR). Only 1 participant in MF group had confirmed PR.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Mycosis Fungoides (MF) | Sezary Syndrome (SS)
Number analyzed (Participants) | 1 | 0
days | 141 [NA to NA] — Only 1 participant was analyzed, therefore actual value was reported and the 95% confidence interval was not applicable. |

3. Secondary Outcome: Time to Progression
Description: Elapsed time from enrollment (baseline) to date of Progressive Disease (PD) as per mSWAT for Mycosis Fungoides (MF) group; mSWAT and Sezary count for Sezary Syndrome (SS) group. mSWAT: weighted sum of percent (%) of total body surface area attributed to skin lesions; scores [0 (unaffected) to 400 (severely affected)] transformed to responses. PD: ≥25% of mSWAT score from nadir. Sezary cells percentage in lymphocytes measured using flow cytometry. PD: ≥40% Sezary cells from nadir. Responders or those who died without PD were censored at the date of the last progression-free disease assessment. Responders who received subsequent systemic anticancer therapy were censored at the date of the last progression-free disease assessment prior to post-discontinuation therapy.
Time Frame: Baseline to measured PD [up to 9 cycles (28-day cycles)]
Population: All participants who received at least 1 dose of study drug. Ten (10) participants were censored for MF group and 2 participants were censored for SS group for this analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Mycosis Fungoides (MF) | Sezary Syndrome (SS)
Number analyzed (Participants) | 19 | 6
days | 78 [50 to 107] | 44 [4 to 82]

4. Secondary Outcome: Time to Objective Response for Responding Participants
Description: Elapsed time from date of study enrollment (baseline) to first evidence of Complete Response (CR) or Partial Response (PR) as per mSWAT for Mycosis Fungoides (MF) group; mSWAT and Sezary count for Sezary Syndrome (SS) group. mSWAT: weighted sum of percent (%) of total body surface area attributed to skin lesions; scores [0 (unaffected) to 400 (severely affected)] transformed into responses. As per mSWAT (CR: No detectable malignant disease for ≥4 weeks. PR: ≥50% mSWAT score reduction from baseline). Sezary cells percentage in lymphocytes measured using flow cytometry. As per Sezary count (CR: Sezary cells <5%; PR: ≥50% reduction in Sezary cells from baseline). Response must be confirmed, but the time to objective response ended at the first assessment. Participants who were not confirmed responders did not contribute to the time to objective response calculation.
Time Frame: Baseline to confirmed response [up to 9 cycles (28-day cycles)]
Population: Participants with confirmed response (CR or PR). Only 1 participant in MF group had confirmed PR.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Mycosis Fungoides (MF) | Sezary Syndrome (SS)
Number analyzed (Participants) | 1 | 0
days | 50 [NA to NA] — Only 1 participant was analyzed, therefore actual value was reported and the 95% confidence interval was not applicable. |

5. Secondary Outcome: European Quality of Life Questionnaire-5 Dimensions (EQ-5D) Health State Utility Score United States (US) Index (Participant-Reported Measure of Health-State Utility)
Description: EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood using a 3-level scale (1 (no problem), 2 (some problems), and 3 (extreme problems)). These combinations of attributes were converted into a single summary health-state index score by applying weights from the US-specific value set to the scoring algorithm. The EQ-5D US value set of health state index scores ranged from 0 (worst imagined health state) to 1 (best imagined health state).
Time Frame: Baseline to study completion [up to 9 cycles (28-day cycles)], end of treatment reported
Population: Enrolled participants who had a baseline and at least 1 post-baseline EQ-5D observation. Last available assessment was reported, last available assessment for a given endpoint defined as efficacy summaries presented as end of study summary.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enzastaurin: Enzastaurin 1125 milligrams (mg) loading dose (total 9 tablets; three 125-mg tablets administered orally 3 times) on Day 1 followed by 500 mg enzastaurin (total 4 tablets; two 125-g) tablets administered orally twice daily) with a minimum of 8 hours between the 2 doses starting on Day 2 until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
Arm/Group | Enzastaurin
Number analyzed (Participants) | 25
units on a scale | 0.7 (0.2)

6. Secondary Outcome: Pruritus 5-Item Severity Assessment Questionnaire (Participant-Reported Experiences With Pruritus)
Description: Participants assessed their present level of itch through the use of an 11-point numeric rating scale anchored at 0 (no itch) and 10 (itch as bad as can be imagined).
Time Frame: Baseline to study completion [up to 9 cycles (28-day cycles)], end of treatment reported
Population: Enrolled participants who had a baseline and at least 1 post-baseline pruritus assessment observation. Last available assessment was reported, last available assessment for a given endpoint defined as efficacy summaries presented as end of study summary.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzastaurin
Number analyzed (Participants) | 25
units on a scale | 5.0 (3.6)

7. Secondary Outcome: Change From Baseline in Itchy Quality of Life (QoL) Domain and Total Scores (Participant-Reported Experiences With Pruritus)
Description: The Itchy QoL is a non-validated 22-item questionnaire designed to assess pruritus-associated symptoms with a 7-day recall using 3 domains: Emotions (9 items), Functions (7 items) and Symptoms domain (6 items). Each Itchy QoL item was evaluated by level of itch frequency through the use of a 5-point adjectival scale 1 (never), 2 (rarely), 3 (sometimes), 4 (often), 5 (all the time). Unweighted means were calculated individually for the 3 domains each with scores range from 1 to 5 and the total score is expressed as the mean of the three dimension scores and ranges from 1 (no itch) to 5 (worst imaginable itch).
Time Frame: Baseline, up to study completion [up to 9 cycles (28-day cycles)], end of treatment reported
Population: Enrolled participants who had a baseline and at least 1 post-baseline Itchy QoL observation. Last available assessment was reported, last available assessment for a given endpoint defined as efficacy summaries presented as end of study summary.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzastaurin
Number analyzed (Participants) | 20
units on a scale
  Symptoms Domain | -0.02 (0.78)
  Emotions Domain | -0.09 (0.63)
  Functions Domain | 0.23 (0.69)
  Total Score | 0.03 (0.59)

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) or Deaths (Safety and Tolerability of Enzastaurin)
Description: Data presented are the number of participants who experienced 1 or more AEs or any serious AEs (SAEs) regardless of causality, deaths during the study including 30 days after treatment discontinuation. A summary of SAEs and other non-SAEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline to study completion [up to 9 cycles (28-day cycles)] plus 30-day safety follow-up
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 25
Participants
  AEs | 20
  SAEs | 5
  Death due to progressive disease | 1

ADVERSE EVENTS:
Description: Study-specific clinical outcomes due to Progressive Disease (PD) were not considered to be a SAE unless the investigator deemed it related to the use of the study drug.
Arm/Group | Enzastaurin
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=25)
Pain (General disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Genital herpes (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Enzastaurin (N=25)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 3 (4)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 6 (6)
Oedema peripheral (General disorders) | 5 (5)
Staphylococcal infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Prostatic pain (Reproductive system and breast disorders) | 1/12 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The study ended at Stage 1 as the minimum level of efficacy was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days